CLINICAL TRIAL: NCT05148533
Title: A Phase I/II Dose Escalation and Expansion Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Efficacy of TJ011133 in Combination With Toripalimab in Subjects With Advanced Solid Tumors
Brief Title: A Study of Single Drug TJ011133 and Toripalimab Combine Treatment for Advanced Solid Tumor
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company Development strategy adjustment
Sponsor: TJ Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ011133STM104
Record Dates: First submitted 2021-11-25; First posted 2021-12-08 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TJ1133 Injection (Experimental)
  Interventions: Drug: TJ1133 Injection

INTERVENTIONS:
Drug: TJ1133 Injection — TJ011133 (30 mg/kg, 45 mg/kg,QW) in combination with toripalimab injection (240 mg, Q3W)

SUMMARY:
This study is a phase I/II study of single drug TJ011133 and Toripalimab combine treatment forAdvanced solid tumor. This study include two stages. First stage is dose escalation and second stage is dose extension. The purpose of part A is to comfirm the MTD or MED and the clinical dose. The purpose of part B is to observe the safty, effectiveness, PK, PD and biomarker properties for effective subjects.

DETAILED DESCRIPTION:
This is an open-label, multi-center phase I/II clinical trial which will enroll 96 to 102 subjects with advanced solid tumors.

This study consists of two phases, the first of which is the dose escalation study of TJ011133 in combination with toripalimab, and the second stage is a dose expansion study.

In phase 1, approximately 3 to 6 subjects will be enrolled in each group to receive TJ011133 (30 mg/kg, 45 mg/kg, QW) in combination with toripalimab injection (240 mg, Q3W). A safety assessment committee, consisting of the sponsor and the investigator, will assess the safety of the first 3 subjects at day 21 after the first dose to determine the safety of the doses as well as to determine whether to enroll 3 additional patients to continue to evaluate the safety.

In the dose expansion phase, patients with melanoma, gastric cancer, and head and neck squamous cell carcinoma will be enrolled, with 30 patients for each malignancy, with a total of 90 patients. TJ011133 will be administered at a prespecified dose of 30 mg/kg or 45 mg/kg, QW or at a less frequency of Q2W or Q3W, and the dosing regimen will be determined based on the safety data obtained by PK/PD model analysis from other TJ011133 clinical studies. And TJ011133 will be given in combination with toripalimab injection at 240 mg, Q3W, until the occurrence of endpoint events such as intolerance or progressive disease.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥18 years old (inclusive);
2. ECOG score: 0-1 points;
3. Patients with histologically or cytologically confirmed locally advanced or metastatic solid tumors, and those who failed or were intolerant to standard therapy, or have no effective treatment options:

   * Enrollment of patients with advanced solid tumors in the dose escalation phase;
   * Subjects with melanoma, gastric cancer, head and neck squamous cell carcinoma will be enrolled in the dose expansion phase;
4. Collect FFPE tumor tissue slides: Collect 12 to 13 archival pre-treatment (mandatory) and 10 on-treatment (optional) paraffin sections from fresh tumor biopsies.
5. Subjects with at least 1 measurable lesion as per RECIST V1.1;
6. Expected survival ≥ 3 months;
7. Main organ function is normal (within 7 days prior to the first dose), i.e., relevant laboratory test criteria are met, and some laboratory indicators meet the following criteria:

   a) Hematology: i. Hemoglobin ≥ 11.0 g/dL or 6.8 mmol/L, received no blood transfusion within 7 days of evaluation, and without dependence on erythropoietin (EPO), ii. Absolute neutrophil count (ANC) ≥1.5×109/L, iii. Platelets ≥ 75×109/L; b) Renal function: i. Creatinine clearance ≥ 45 mL/min (calculated by Cockcroft-Gault formula), ii. Qualitative urine protein ≤ 1+; or qualitative urine protein ≥ 2+, 24-hour urine protein < 1 g; c) Liver function i. Serum total bilirubin ≤ 1.5 × ULN, ii. Both aspartate aminotransferase (AST, SGOT) and alanine aminotransferase (ALT, SGPT) ≤ 2.5 × ULN, iii. Serum albumin ≥ 2.8 g/dL (received no albumin infusion within 2 weeks prior to blood collection); d) Coagulation function: i. International normalized ratio (INR), or prothrombin time (PT) ≤ 1.5 x ULN, or PT parameters can be maintained ≤ 1.5 x ULN with an anticoagulant at a stable dose, ii. Activated partial thrombin time (aPTT) ≤ 1.5 × ULN, or aPTT parameters can be maintained ≤ 1.5 × ULN with the use of anticoagulants;
8. Male subjects with reproductive potential and female subjects with pregnancy potential (which refer to men or women who have not been surgically sterilized, and women who are not post-menopausal) must use highly effective contraceptive methods such as oral contraceptives, intrauterine devices, sexual abstinence or barrier contraception in conjunction with spermicides during the course of the study and until 6 months after the last dose;
9. Subjects who are willing to participate in this study and sign the ICF, have good compliance and cooperate with the follow-up.

Subjects must be excluded if they meet any of the following criteria:

1. Pregnant or breast-feeding women;
2. Have received prior treatment with CD47 or SIRPα inhibitors;
3. Have received prior treatment with CAR-T cell therapy;
4. Have received systemic anti-tumor therapy within 4 weeks prior to the start of the study treatment, except for the following;

   * Have received nitrosoureas or mitomycin C within 6 weeks prior to the first dose of the investigational product;
   * Have received oral fluorouracils and small-molecule targeted agents within 2 weeks prior to the first dose of the investigational product or within 5 half-lives of the drug, whichever is longer;
   * Have received traditional Chinese medicine with anti-tumor indications within 2 weeks prior to the first dose of the investigational product.
5. With present or previous history of two or more primary tumors, except for cured carcinoma in situ and basal cell carcinoma. Subjects with concurrent tumors that have remained stable for more than 5 years prior to study enrollment are eligible;
6. Subjects who have active auto-immune diseases requiring systemic treatment with immunomodulatory drugs within 12 months prior to treatment initiation, but relevant alternative therapies are allowed;
7. Subjects who have received systemic treatment with corticosteroids (at doses higher than 10 mg/day prednisone or the equivalent) or other immunosuppressants for more than 7 days within 2 weeks prior to the start of the study treatment (use of inhaled or topical steroids or an adrenal replacement therapy at a dose exceeding 10 mg prednisone equivalents is acceptable in the absence of active auto-immune diseases);
8. Subjects who have received other unmarketed investigational drugs or treatment within 4 weeks prior to the start of the study treatment;
9. Subjects who have undergone major surgeries or were severely traumatized within 4 weeks prior to the start of the study treatment, or those who are recovering from such surgeries or traumas and the study results will be affected in the opinion of the investigator, or those have been scheduled to undergo surgeries during their participation in the study;
10. Have received chest radiotherapy or extended field radiotherapy (defined as more than 50% pelvic bone mass or equivalent) within 4 weeks prior to the initiation of study treatment, or palliative radiotherapy within 2 weeks prior to the initiation of treatment;
11. With the presence of symptomatic central nervous system (CNS) metastases and neurological instability or a need to increase the dose of corticosteroids to control CNS symptoms within 2 weeks prior to the start of the study treatment;
12. Have positive HBsAg and HBV-DNA > 500 IU/mL or the lower limit of detection of the study site [only if the lower limit of detection at the site is higher than 500 IU/mL]); HCV antibody positive and HCV-RNA quantitative detection is above the upper limit of normal;
13. With known positive human immunodeficiency virus (HIV) serum reaction;
14. With uncontrolled hydrothorax, ascites, or pericardial effusion;
15. Subjects who have or had prior active interstitial lung disease;
16. Subjects with hypertension that cannot be well controlled with drug therapies. Clinical uncontrollable hypertension is defined as a systolic blood pressure > 150 mm Hg or a diastolic blood pressure > 90 mm Hg (adjustment of anti-hypertensive drugs before the start of this study is acceptable, but the average blood pressure of the most recent three consecutive recordings must ≤ 150/90 mm Hg prior to enrollment of the study);
17. Adverse reactions to prior anti-tumor therapy have not recovered to Grade ≤ 1 as per CTCAE Ver 5.0 (except for toxicities that are judged by the investigator to have no safety risk, such as alopecia, Grade 2 peripheral neurotoxicity, hypothyroidism which is stable after hormone replacement therapy, etc.);
18. Have received immunotherapy and experienced Grade ≥ 3 irAEs or Grade ≥ 2 immune-related myocarditis;
19. Subjects with clinically significant cardiovascular disorder: including Grade II to IV cardiac insufficiency defined by the classification criteria of New York Heart Association (NYHA), congestive cardiac failure, heart block above Grade II, infarct myocardial within the past 3 months, unstable arrhythmia or unstable angina, significant QT interval prolongation (>450 ms for male and >470 ms for female); or cerebral infarction within the past 3 months, or surgical history of percutaneous transluminal coronary angioplasty (PTCA) or coronary artery bypass grafting (CABG) within the past 6 months;
20. With deep vein thrombosis within 6 months prior to the start of study treatment (except for the subjects who have not used the anti-coagulation agent of warfarin for more than 2 weeks prior to the start of the study treatment);
21. Thrombolytic therapy (except for the maintenance of an IV catheter) within 10 days prior to treatment initiation;
22. Any active infection requiring intravenous anti-infective therapy;
23. Subjects with known or suspected conditions (e.g., alcoholism, drug dependence, or psychological disorder) which render it impossible for them to comply with the protocol, or who may be at rick if they participate in this study according to the opinion of the investigator; or with the conditions in which subject's participation in this study is not their best option as judged by the investigator, (e.g., causing harm to health) or that affect, limit, or confound protocol assessments.

Exclusion Criteria:

1. Pregnant or breast-feeding women;
2. Prior treatment with CD47 or SIRPα inhibitors;
3. Prior CAR-T cell therapy;
4. Subjects who have received systemic anti-tumor therapies within 4 weeks prior to the initiation of treatment or within five half-lives (whichever is shorter) of the study drug, except for the following;

   * Nitrosourea or mitomycin C within 6 weeks prior to the first dose of study drug;
   * Oral fluorouracils and small molecule targeted agents are within 2 weeks prior to the first dose of study drug or within 5 half-lives of the drug, whichever is longer;
   * Traditional Chinese medicine with anti-tumor indications is within 2 weeks prior to the first dose of study drug.
5. Subjects who had or have two or more primary tumors cannot be enrolled, except for cured carcinoma in situ and basal cell carcinoma. Subjects with concomitant tumors that have been stable for more than 5 years before enrollment in the study can be enrolled;
6. Subjects who have active auto-immune diseases requiring systemic treatment with immunomodulatory drugs within 12 months prior to treatment initiation, but relevant alternative therapies are allowed;
7. Subjects who have received systemic treatment with corticosteroids (more than 10 mg/day prednisone equivalent) or other immunosuppressants for more than 7 days within 2 weeks prior to treatment initiation (inhaled or topical steroids or adrenal replacement therapy in excess of 10 mg prednisone equivalents is permitted in the absence of active auto-immune disease);
8. Subjects who have participated in clinical trials (including investigational vaccines), and received interventional and investigational treatment with invasive and investigational medical devices within 4 weeks prior to the initiation of treatment;
9. Subjects who have experienced major surgery or severe trauma within 4 weeks prior to treatment initiation, or who are recovering, but which will exert an impact on the study as judged by the investigator, or who have surgical arrangements during their participation in the study;
10. Chest radiotherapy or expanded field radiotherapy (defined as more than 50% pelvic bone mass or equivalent) within 4 weeks prior to the initiation of treatment, or palliative radiotherapy within 2 weeks prior to the initiation of treatment;
11. Presence of symptomatic metastases to the central nervous system (CNS) and neurological instability within 2 weeks prior to initiation of dosing or a need to increase the dose of steroids to control CNS symptoms;
12. HBsAg positive and HBV-DNA copies > 500 IU/ml or lower limit of detection at the site (only if the lower limit of detection at the site is above 500 IU/ml); HCV antibody positive and result of HCV-RNA quantitative assay above the ULN;
13. Known positive human immunodeficiency virus (HIV) serum reaction;
14. Subjects with uncontrollable hydrothorax, ascites, or pericardial effusion;
15. Subjects who have or had active interstitial lung disease;
16. Subjects with hypertension that cannot be well controlled with drug therapies. Hypertension which cannot be controlled clinically is defined as a systolic blood pressure > 150 mmHg or a diastolic blood pressure > 90 mmHg (adjustment of treatment medications for hypertension is allowed before the initiation of this study, but the average blood pressure calculated from the most recent three consecutive recordings must ≤ 150/90 mmHg prior to his/her entry into the study);
17. Adverse reactions of prior anti-tumor therapy have not recovered to ≤ CTCAE 5.0 Grade 1 (except for alopecia, Grade 2 peripheral neurotoxicity and other toxicities judged by the investigator to have no safety risk);
18. Subjects with clinically significant cardiovascular disorder: including Grade II to IV cardiac insufficiency defined by the classification criteria of New York Heart Association (NYHA), congestive cardiac failure, heart block above Grade II, infarct myocardial within the past 3 months, unstable arrhythmia or unstable angina, significant QT interval prolongation (>450 ms for male and >470 ms for female); or cerebral infarction within the past 3 months, or surgical history of percutaneous transluminal coronary angioplasty (PTCA) or coronary artery bypass grafting (CABG) within the past 6 months;
19. Deep vein thrombosis within 6 months prior to the initiation of treatment (except for the case where warfarin has not been used for anti-coagulation for more than 2 weeks prior to treatment initiation);
20. Thrombolytic therapy (except for the maintenance of an IV catheter) within 10 days prior to treatment initiation;
21. Any active infection requiring intravenous anti-infective treatment;
22. Subjects with known or suspected conditions (e.g., alcoholism, drug dependence, or psychological disorder) which render it impossible for them to comply with the protocol, or who may be at risk if they participate in this study according to the opinion of the investigator; or with the conditions in which subject's participation in this study is not their best option as judged by the investigator, (e.g., causing harm to health) or that affect, limit, or confound protocol assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Incidence and Severity of Adverse Events | throughout the dose escalation assessed to 1year
  The NCI CTCAE V5.0 will be used to assess adverse events on this study
The Objective Response Rate(ORR) | Through the dose expansion assessed to 1 year
  The Objective response rate will be assessed by RECIST v1.1 criteria in this study.

CONTACTS AND LOCATIONS:
Locations (22):
- China (22):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Province Cancer Hospital, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Guangzhou Medical University Affiliated Tumor Hospital, Guangzhou, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University Of Science And Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - HuNan Cancer Hospital, Changsha, Hunan
  - The first affiliated hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shandong Tumor Hospital, Jinan, Shandong
  - Shanghai Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang